CLINICAL TRIAL: NCT00412685
Title: Quantification of the Myocardial Microcirculation by Contrast Echocardiography In Adult Patients With Congenital Heart Disease
Brief Title: Myocardial Contrast Echocardiography in Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Christian Seiler, MD, Professor and Co-Chairman of Cardiology, Department of Cardiology, University Hospital, CH-3010 Bern, Switzerland
Other Study IDs: 70/06
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: D-Transposition of Great Arteries; Tetralogy of Fallot
MeSH Terms: conditions — Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- TGA group: The TGA group consists of 15 patients treated withMustard or Senning procedures for surgical repaired of D-TGA atrial switch operation.
- TOF group: The TOF group consists of 15 patients with surgically corrected TOF.
- Control group: The control group C consists of 15 control subjects (AH) with normal Doppler Echocardiographic echocardiographic examinations.

SUMMARY:
Patients with congenital heart disease in whom the right ventricle is exposed to pressure or volume overload show progressive systolic dysfunction of the right ventricle, the fact of which conveys substantial morbidity and mortality. The aim of this study is to investigate the myocardial perfusion in these patients by myocardial contrast echocardiography (MCE) in order to determine whether disturbed blood flow plays a role in the development of right ventricular systolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* D-TGA or Fallot-Tetralogy or Healthy person
* written informed consent
* Age >= 18 years

Exclusion Criteria:

* Anaemia
* Pregnancy and breast feeding
* Diabetes mellitus
* Contraindications to stress testing (ergometry or adenosine)
* Known adverse reaction or hypersensitivity against V08DA (SonoVue) or its components or against adenosine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is divided in three groups, which are all age- and gender-matched. The TGA group consists of 15 patients treated withMustard or Senning procedures for surgical repaired of D-TGA atrial switch operation. The TOF group consists of 15 patients with surgically corrected TOF. The control group C consists of 15 control subjects (AH) with normal Doppler Echocardiographic echocardiographic examinations.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2006-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Seiler, Prof., Principal Investigator — University Hospital Berne, Switzerland
Locations (1):
- University Hospital Inselspital, Bern, Switzerland